CLINICAL TRIAL: NCT01107028
Title: Pulmonary Rehabilitation for Idiopathic Pulmonary Fibrosis
Brief Title: Beneficial Effects of Pulmonary Rehabilitation for Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NJ230; K23HL092227-01A2 (NIH)
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; Dyspnea; Functional capacity; Quality of life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rehab: Subjects randomized to the Rehab group will have data collected at baseline and then within one week enroll in a pulmonary rehabilitation program. Data will again be collected within one week of completing pulmonary rehabilitation and again six months later.
  Interventions: Other: Standard pulmonary rehabilitation program
- Wait: Subjects randomized to the Wait group will have data collected at baseline and wait eight weeks before enrolling in a pulmonary rehabilitation program. Data will again be collected within one week of completing pulmonary rehabilitation and again six months later.
  Interventions: Other: Standard pulmonary rehabilitation program

INTERVENTIONS:
Other: Standard pulmonary rehabilitation program — At the assigned time, subjects will complete a six-week, outpatient pulmonary rehabilitation program at any local center that has such a program.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a devastating disease marked by progressive lung scarring leading to multiple life-altering sequelae. The over-arching goals of the principal investigator's research program are to more fully characterize these sequelae and to examine interventions that might improve them. The hypotheses of this particular study are that pulmonary rehabilitation (PR) is one such intervention, and that PR will improve the sequelae of dyspnea and impairments in functional capacity, cognition, mood and anxiety, fatigue, and quality of life (QOL) in patients with IPF.

DETAILED DESCRIPTION:
Subjects will come to our center to be enrolled. Baseline data collection (performance of a six-minute walk test and completion of questionnaires) and randomization to one of two groups--either Rehab or Wait--will take place at the same enrollment visit if time permits. Subjects in either group will complete pulmonary rehabilitation, just at slightly different times, depending on which group they are randomized to.

Pulmonary rehabilitation is a program run by respiratory and/or physical therapists and other health professionals that involves exercise, education, and support with the goals to improve functional capacity, symptom management, and well-being. It will last 6-8 weeks, during which time, subjects will complete 18 approximately hour-long sessions. Pulmonary rehabilitation may be completed at any local center that makes travel convenient.

Data collection visits will take place at National Jewish Health at baseline, eight weeks (without intervening pulmonary rehabilitation in the Wait group), after completion of pulmonary rehabilitation (time varies, depending on the randomization group), and finally six months after completion of the pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* IPF
* Able to walk unassisted for balance
* Able to speak and understand English well enough to complete complex tasks with directions given in English

Exclusion Criteria:

* Pulmonary fibrosis not due to IPF
* Coexisting comorbid conditions that would make exercise contraindicated

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic pulmonary fibrosis, as defined by the American Thoracic Society Consensus Guidelines
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Six-minute walk distance | Eight weeks
  Distance walked during a standard six-minute walk test.

SECONDARY OUTCOMES:
dyspnea, fatigue, anxiety, depression, quality of life | Eight weeks
Six minute walk distance | Six months after completion of pulmonary rehabilitation
dyspnea, fatigue, anxiety, depression, quality of life | Six months after completion of pulmonary rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Swigris, DO, MS, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Swigris JJ, Brown KK, Make BJ, Wamboldt FS. Pulmonary rehabilitation in idiopathic pulmonary fibrosis: a call for continued investigation. Respir Med. 2008 Dec;102(12):1675-80. doi: 10.1016/j.rmed.2008.08.014. Epub 2008 Oct 10. PMID 18848771